CLINICAL TRIAL: NCT04474353
Title: A Phase 1 Study of Tumor Treating Fields With 5 Day Hypofractionated Stereotactic Radiosurgery and Concurrent and Maintenance Temozolomide in Newly Diagnosed Glioblastoma
Brief Title: Study of Tumor Treating Fields With Hypofractionated Chemoradiotherapy in Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Principal Investigator, Scott Soltys, Professor of Radiation Oncology (Radiation Therapy), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-53582; NCI-2021-06752 (Other: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma; Newly Diagnosed Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Gadolinium; Contrast Media; Temozolomide; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Novo-TTF (Experimental): Day 1: Subjects will wear the Optune (TTFields device) for ≥ 18 hours/day. They will take off the device when receiving stereotactic radiosurgery and brain MRI scans.
  Days 1 to 8: Subjects will take oral temozolomide 75 mg/m2/day Days 2 to 8: Subjects will receive stereotactic radiosurgery (total of 35 Gy) divided equally over 5 days
  • After the interventional treatment, subjects will receive standard of care adjuvant chemotherapy and routine surveillance brain MRI scans.
  Interventions: Device: Optune; Drug: Gadolinium; Drug: Temozolomide; Radiation: Stereotactic radiosurgery (SRS)

INTERVENTIONS:
Device: Optune — Noninvasive, portable device which generates tumor treating fields (TTFields) manufactured by Novocure
Drug: Gadolinium — Gadolinium contrast medium
  Other Names: Contrast agent
Drug: Temozolomide — Chemotherapy agent
Radiation: Stereotactic radiosurgery (SRS) — Standard of Care: SRS (35 Gy in 5 fractions of 7 Gy), 5-day treatment from Day 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the combination therapy of TTFields + SRS+ Temozolomide (TMZ) for newly diagnosed glioblastoma (GBM).

DETAILED DESCRIPTION:
Primary Objective:

Determine the safety of Tumor Treating Fields (TTFields) started concurrently with 5 fraction stereotactic radiosurgery (SRS) and temozolomide for newly diagnosed glioblastoma. secondary objective: Efficacy for the combination of TTFields started concurrently with 5

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven newly diagnosed glioblastoma (GBM, WHO Grade IV) or molecular GBM of lower grade that will be treated as per glioblastoma (defined as IDH wild type, 1p19q not co deleted)
* Age ≥ 18 years
* A maximum tumor target diameter of less than 5 cm on the post operative MRI used for SRS planning (a 5 mm margin is added in the radiotherapy planning process, yielding a maximum diameter of the planning target volume (PTV) of less than 6 cm). If the maximum diameter is greater than 5 cm, the subject is still eligible if the PTV is less than 113 cm3 which is the volume of a 6 cm diameter sphere.
* Adequate organ function (obtained within 14 days prior to Day 0) as evidenced by:

  * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L without myeloid growth factor support for 7 days preceding the lab assessment
  * Hemoglobin (Hgb) ≥ 9 g/dL (90 g/L); < 9 g/dL (< 90 g/L) is acceptable if hemoglobin is corrected to ≥ 9 g/dL (90 g/L) as by growth factor or transfusion prior to Day 0
  * Platelet count ≥ 100 × 109/L without blood transfusions for 7 days preceding the lab assessment
  * Bilirubin ≤ 1.5 × upper limit of normal (ULN), except for subjects with documented history of Gilbert's disease
  * Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 2.5 × ULN
  * Alkaline phosphatase (AP) ≤ 3 × ULN
  * Women of childbearing potential (WCBP): negative serum pregnancy test (this test is required of all women unless post menopausal, defined as 12 consecutive months since last regular menses or surgically sterile)
* Ability to tolerate MRI
* Karnofsky Performance Scale (KPS) ≥ 60
* Ability to understand and the willingness to sign (personally or by a legal authorized representative) the written IRB approved informed consent document.

Exclusion Criteria:

* Previous chemotherapy or radiotherapy for glioma
* Concurrent use of experimental therapies
* Known allergy to adhesive tapes or other skin adhesives used in medical care
* Known underlying skin hypersensitivity or other condition of the scalp with potential toxicity per pre treatment dermatology evaluation
* Subjects with the following co morbid disease or incurrent illness:

  * Subjects with known cirrhosis diagnosed with Child Pugh Class A or higher liver disease.
  * Prior malignancy except for non melanoma skin cancer and carcinoma in situ (of the cervix or bladder), unless diagnosed and definitively treated more than 3 years prior to first dose of investigational drug
  * Severe/uncontrolled inter current illness within the previous 28 days prior to first day of treatment
  * Subjects who have implantable devices that are contra indicated for use with TTFields
  * Any other significant co morbid conditions that in the opinion of the investigator would impair study participation or cooperation.
* Subjects receiving the following medications at the time of combined TTFields and SRS:

  * Pharmacotherapy for tuberculosis or HIV as these medications are known to interact with temozolomide
  * Other chemotherapy, other investigational agents, or biologic agents for the treatment of cancer including antibodies (eg, bevacizumab, trastuzumab, pertuzumab), small molecules, or any investigational agent(s).
* Pregnant or nursing females will be excluded from the study
* History of inability to tolerate MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLTs) | 5 months
  Dose limiting toxicities (DLTs) are defined as possibly, probably, or definitely related adverse events that are severe or medically significant, and needing topical & systemic therapy; needing surgery intervention; needing hospitalization; needing treatment interruption; or life threatening. Late DLTs will be assessed as the number of DLTs that occur in the period from 31 days after the start of treatment through 5 months after the start of treatment. The outcome will be reported as a number without dispersion.

SECONDARY OUTCOMES:
Acute dose limiting toxicity | 1 month
  Dose limiting toxicities (DLTs) are defined as possibly, probably, or definitely related adverse events that are severe or medically significant, and needing topical & systemic therapy; needing surgery intervention; needing hospitalization; needing treatment interruption; or life threatening. Acute DLTs will be assessed as the number of DLTs that occur in the period from the start of treatment through 30 days after the start of treatment. The outcome will be reported as a number without dispersion.
Progression-free Survival (PFS) at 6 Months | 6 months
  Progression-free survival is defined as the number of evaluable participants who, at 6 months from the date of surgical resection or biopsy (PFS6), are alive without disease progression, death, or other defined event (study withdrawal or loss to follow up). Disease progression is defined as ≥ 25% increase in product of perpendicular diameters of the lesion; any increase in MRI T2/FLAIR lesion area from previous MRI scan; MRI detection of a new lesion; decline in clinical status not attributable to causes other than the tumor. The outcome will be reported as the number without dispersion.
Overall Survival (OS) | 30 months
  Overall survival (OS) will be assessed as the number of evaluable participants who remain alive from the date of surgical resection or biopsy. The outcome will be reported as the number without dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Scott G Soltys, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No